CLINICAL TRIAL: NCT02624128
Title: Preclinical and Clinical Study of Valproic Acid Plus Cisplatin and Cetuximab in Recurrent and/or Metastatic Squamous Cell Carcinoma of Head and Neck
Brief Title: Valproic Acid Plus Cisplatin and Cetuximab in Recurrent and/or Metastatic Squamous Cell Carcinoma of Head and Neck
Acronym: V-CHANCE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V-CHANCE; 2014-001523-69 (EudraCT Number)
Record Dates: First submitted 2015-11-26; First posted 2015-12-08 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: head and neck cancer; valproic acid; recurrent; metastatic
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Valproic Acid; Cisplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- valproic acid plus cisplatin and cetuximab (Experimental)
  Interventions: Drug: Valproic Acid; Drug: Cisplatin; Drug: Cetuximab

INTERVENTIONS:
Drug: Valproic Acid — Treatment will be administered orally starting at day -14, with 500 mg slow releasing tablet at evening. Thereafter, the dose will be increased also using 300 mg tablets until reaching 1500 mg on day -1. The titration strategy is to reach a target VPA serum level of 50-100 μg/ml.
Drug: Cisplatin — administered intravenously at dose of 75 mg/m2 given every three weeks for 6 cycles
Drug: Cetuximab — administered intravenously at induction dose of 400 mg/m2 followed by maintenance doses of 250 mg/m2 given weekly

SUMMARY:
V-CHANCE is a phase 2, trial exploring the feasibility and the activity of valproic acid (VPA) in combination with the standard cisplatin-cetuximab combination in patients with recurrent/metastatic squamous cell carcinoma of the head and neck, never treated with first-line chemotherapy. The study includes an explorative analysis of the potential prognostic or predictive role of several biomarkers with the aim of improving the knowledge of the mechanisms by which VPA enhances chemotherapy effect and of identifying early predictors of treatment response/resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven squamous cell carcinoma of head and neck with exclusion of the nasopharynx
2. First-line recurrent and/or metastatic disease
3. No prior chemotherapy except for chemoradiation or induction chemotherapy followed by local treatment given in the context of a curative strategy.
4. age> 18 years
5. ECOG Performance Status ≤1
6. Life expectancy at least 3 months at study entrance
7. Normal bone marrow reserve (absolute neutrophil count > 1500/mm3; platelets > 100000/mm3; haemoglobin> 9 g/dl)
8. Normal hepatic function (total serum bilirubin < 1.5 x upper limit of normal; liver transaminases < 3 x upper limit of normal)
9. Normal renal function (serum creatinine < 1,25 x upper limit of normal and creatinine clearance > 60 ml/min).
10. Normal cardiac function (assessed by ECG and echocardiography with ejection fraction > 50%)
11. Effective contraception for both male and female patients if the risk of conception exist
12. Signed written informed consent

Exclusion Criteria:

1. Concomitant treatment with other experimental drugs.
2. Brain metastases (CT scan or MRI required only in case of clinical suspicion of CNS metastases)
3. Non squamous cell histology
4. Any concurrent malignancy. Patient with a previous malignancy but without evidence of disease for 5 years will be allowed to enter the trial.
5. History of myocardial infarction within the last 12 months
6. ECOG PS ≥ 2
7. Significant cardiovascular comorbidity (e.g. myocardial infarction, superior vena cava [SVC] syndrome, patients with an ejection fraction of <50%) or presence of cardiac disease that in the opinion of the Investigator increases the risk of ventricular arrhythmia.
8. History of arrhythmia (multifocal premature ventricular contractions [PVCs], bigeminy, trigeminy, ventricular tachycardia, or uncontrolled atrial fibrillation) which is symptomatic or requires treatment (CTCAE grade 3) or asymptomatic sustained ventricular tachycardia. Patients with long QT-syndrome or QTc interval duration > 480 msec or concomitant medication with drugs prolonging QTc.
9. HIV positive patients
10. Patients who cannot take oral medication, who require intravenous feeding, have had prior surgical procedures affecting absorption, or have active peptic ulcer disease.
11. Known or suspected hypersensitivity to any of the study drugs.
12. Patients who have had prior treatment with an HDAC inhibitor and patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid.
13. Major surgical procedure within 28 days prior to study treatment start.
14. Pregnant or lactating women.
15. Women of childbearing potential with either a positive or no pregnancy test at baseline (postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential)l.
16. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2015-02-23 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with an objective response | up to 4 years
  Response will be assessed according to RECIST v1.1 criteria

SECONDARY OUTCOMES:
overall survival | up to 6 years
time to tumor progression | up to 6 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Caponigro, M.D, Principal Investigator — National Cancer Institute, Naples; Alfredo Budillon, M.D, Principal Investigator — National Cancer Institute, Naples
Locations (1):
- Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Italy

REFERENCES:
- [Derived] Caponigro F, Di Gennaro E, Ionna F, Longo F, Aversa C, Pavone E, Maglione MG, Di Marzo M, Muto P, Cavalcanti E, Petrillo A, Sandomenico F, Maiolino P, D'Aniello R, Botti G, De Cecio R, Losito NS, Scala S, Trotta A, Zotti AI, Bruzzese F, Daponte A, Calogero E, Montano M, Pontone M, De Feo G, Perri F, Budillon A. Phase II clinical study of valproic acid plus cisplatin and cetuximab in recurrent and/or metastatic squamous cell carcinoma of Head and Neck-V-CHANCE trial. BMC Cancer. 2016 Nov 25;16(1):918. doi: 10.1186/s12885-016-2957-y. PMID 27884140